CLINICAL TRIAL: NCT03119545
Title: A Family-Centered Intervention When a Parent is Cared for in Specialized Homecare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Sköndal University College (Other)
Responsible Party: Principal Investigator, Malin Lövgren, Associate professor, Ersta Sköndal University College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/7-31/1
Record Dates: First submitted 2017-04-03; First posted 2017-04-18 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Palliative Care
Keywords: intervention; support program; family centered; parental death
MeSH Terms: conditions — Parental Death

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beardslee family centered intervention (Experimental): This Group will have the family centered program.
  Interventions: Behavioral: Beardslee family centered intervention
- Comparison group (No Intervention): This Group will have standard care

INTERVENTIONS:
Behavioral: Beardslee family centered intervention — The method entails six meetings. The time for the meeting is 1-2 hours and is usually held once per week. Meetings 1 and 2) include only the parents and focus firstly on the ill parent's history and secondly on the well parent/relative. Meeting 3) includes interviews with each child aged 6-19 years, without the parents being present, concerning the child´s understanding of the disease, potential worries and questions. During the interview the child can formulate his or her own questions for the family meeting. Meeting 4) includes the parents and focuses on the planning of the family meeting. The child's thoughts and questions serve as a guide for the upcoming family meeting. Meeting 5) is the family meeting. Meeting 6) is a follow-up with all of the family members.
  Other Names: the family talk intervention
  Arms: Beardslee family centered intervention

SUMMARY:
The overall purpose of this project is to evaluate a family-centered intervention (the Family Talk Intervention, by W. Beardslee) in families where a parent of children aged 6-19 years is seriously ill and cared for in specialized homecare. The aims of the intervention are to increase family communication, the families' awareness of the impending death and their knowledge about the cancer illness, and thereby reduce the family members' long-term psychological distress.

DETAILED DESCRIPTION:
The death of a parent is one of the most traumatic events that can happen to a Child. In our previous research, we have found that a lack of medical knowledge, communication and awareness of impending death increased long-term psychological morbidity among bereaved family members. Unfortunately, very few clinical interventions in palliative care have been conducted in Sweden.There is therefore a need to develop and evaluate interventions that aim to decrease the risk for psychological morbidity in families affected loss.

The overall purpose of this project is to evaluate a family-centered intervention (the Family Talk Intervention, by W. Beardslee) in families where a parent of children aged 6-19 years is seriously ill and cared for in specialized homecare. The aims of the intervention are to increase family communication, the families' awareness of the impending death and their knowledge about the cancer illness, and thereby reduce the family members' long-term psychological distress.

This study is a family-based intervention study among families where a parent of young children is seriously ill. It involves an intervention group and a comparison group. The two groups will consist of families where the seriously ill parent has at least one child in the age range 6-19 years. Around thirty families will be recruited by two interventionists through two specialized homecare unit in Stockholm and this is expected to take about 18 months. Families in the comparison group (N=30) will be recruited by a research member at two other specialized homecare units in the Stockholm area.

The effect of the intervention will be measured by questionnaires to both parents and children. Questionnaire data collection will be conducted before the intervention is started (baseline, for both intervention and control group). After two months there will be a follow-up for both groups. The next follow-up for both groups will be performed one year after the baseline.

In order to examine the meaning of the intervention for all family members and the study-feasibility we are planning to conduct interviews after meeting 5. Interviews with the whole family respectively each family members will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* At least one Child in the family 6-19 years
* Speaking and understanding Swedish
* One parent with severe illness or dying

Exclusion Criteria:

* If the family is in need of interpreter

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Self-reported family communication, change over time | Baseline (start of intervention), follow up 1 (after two months), follow up 2 (after one year).
  Will be measured using study specific questionnaires (6-7 years 26 items; 8-12 years 28 items; 13-19 years 52 items; patient 45 items; parent/other significant adult 54 items).
Self-reported family communication | After five weeks from the start of the intervention
  Will be measured by interviews

SECONDARY OUTCOMES:
Self -reported knowledge about the illness, change over time | Baseline (start of intervention), follow up 1 (after two months), follow up 2 (after one year).
  Will be measured using study specific questionnaires (6-7 years 26 items; 8-12 years 28 items; 13-19 years 52 items; patient 45 items; parent/other significant adult 54 items).
Self -reported knowledge about the illness | After five weeks from the start of the intervention
  will be measured by interviews
Self-reported psychological distress, change over time | Baseline (start of intervention), follow up 1 (after two months), follow up 2 (after one year).
  Will be measured using questionnaires "The pediatric quality of Life inventory" (PEDS QL) (6-7 years 15 items; 8-19 years 16 items). "Generalized Anxiety Disorder Assessment" (GAD-7) for the adults (8 items).

CONTACTS AND LOCATIONS:
Overall Officials: Malin Lövgren, PhD, Principal Investigator — Ersta Sköndal Bräcke University College
Locations (1):
- Ersta Sköndal Bräcke University College, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weber Falk M, Eklund R, Kreicbergs U, Alvariza A, Lovgren M. Breaking the silence about illness and death: Potential effects of a pilot study of the family talk intervention when a parent with dependent children receives specialized palliative home care. Palliat Support Care. 2022 Aug;20(4):512-518. doi: 10.1017/S1478951521001322. PMID 35876452
- [Derived] Eklund R, Alvariza A, Kreicbergs U, Jalmsell L, Lovgren M. The family talk intervention for families when a parent is cared for in palliative care - potential effects from minor children's perspectives. BMC Palliat Care. 2020 Apr 16;19(1):50. doi: 10.1186/s12904-020-00551-y. PMID 32299420
- [Derived] Eklund R, Kreicbergs U, Alvariza A, Lovgren M. The family talk intervention in palliative care: a study protocol. BMC Palliat Care. 2018 Feb 23;17(1):35. doi: 10.1186/s12904-018-0290-8. PMID 29471826